CLINICAL TRIAL: NCT00670813
Title: Verstärkung Der Therapeutischen Wirkung Von Schlafentzug Durch Modafinil - Eine Doppelblinde, Randomisierte, Placebokontrollierte Monozentrische Studie Der Phase II (Enhancing the Therapeutic Efficacy of Sleep Deprivation by Modafinil - a Double Blind, Placebo-controlled Monocentric Phase II Study)
Brief Title: Enhancing the Therapeutic Efficacy of Sleep Deprivation by Modafinil
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Michael H. Wiegand, Professor Dr.med. Dr.med.habil. Dipl.-Psych., Sleep Laboratory Department of Psychiatry and Psychotherapy of the Technical University Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SE03; EudraCT Nr. 2005-003196-21
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2008-04

CONDITIONS: Depression
Keywords: Depression; (total) sleep deprivation; Modafinil; polysomnography sleep
MeSH Terms: conditions — Depression; Sleep Deprivation | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Vigil) (Experimental): "Modafinil" Arm: during the 40 h sleep deprivation period (morning until evening next day) the depressed patient receives 200 mg of Modafinil each at 12:00, 24:00 and again at 12:00 o' clock
  Interventions: Drug: Modafinil (Vigil)
- Placebo (Placebo Comparator): "Placebo" Arm: during the 40 h sleep deprivation period (morning until evening next day) the depressed patient receives Placebo at 12:00, 24:00 and again at 12:00 o' clock
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil (Vigil) — Oral application of 2 x 100 mg Modafinil each encapsulated in identical looking gelatine capsules at 12:00, 24:00 and again at 12:00 o' clock during the 40 h sleep deprivation period
  Arms: Modafinil (Vigil)
Drug: Placebo — Oral application of 2 x 100 mg Placebo each encapsulated in identical looking gelatine capsules at 12:00, 24:00 and again at 12:00 o' clock during the 40 h sleep deprivation period
  Arms: Placebo

SUMMARY:
The study aims to investigate whether the administration of the stimulant modafinil during a 40 hour sleep deprivation period in depressed patients can intensify the antidepressant effect of the sleep deprivation as assessed by a reduction in the Hamilton Depression score (HAMD, 6-item version). We postulate that this also correlates with a reduction of the polysomnographically assessed overall amount of sleep during this period.

DETAILED DESCRIPTION:
In about 60 % of depressed patients, sleep deprivation has an acute therapeutic effect. The effect appears within very few hours; this is different from all other antidepressant treatments. However, in most cases patients relapse after the subsequent night's sleep (Wu & Bunney 1990).

The antidepressant mechanism of action of sleep deprivation is not known as yet; several hypotheses are presented and discussed in various review articles (Wiegand 1995; Kasper & Möller 1996; Wirz-Justice & van den Hoofdakker 1999; Gillin et al. 2001; Ringel & Szuba 2001; Giedke & Schwärzler 2002). At present, the following general hypotheses are most discussed:

1. Sleep deprivation exerts its effect by activating or intensifying an antidepressant "pro-cess". This "process" may be dopaminergic or serotonergic transmission, thyroid function etc.
2. Sleep deprivation inactivates a hypothetic "depressiogenic" substance which is produced during sleep.
3. Sleep deprivation reduces the central nervous cholinergic transmitter activity and restores the balance between cholinergic and aminergic transmitter systems.
4. Sleep deprivation acts by preventing sleep during a "critical" or "vulnerable" phase of circadian rhythms; there are various chronobiological assumptions which can specify such a "critical phase".

Several studies tried to indentify predictors of response to sleep deprivation in order to clarify the mechanism of action. Among clinical predictors is a symptom pattern with "endogenous" or "melancholic" traits and the presence of pronounced diurnal variations of mood, and a behaviour pattern pointing to an elevated level of arousal or activity. Another predictor is a pronounced sleep disturbance during the baseline night. Among the many neuroendocrine and neurohumoral factors which have been studied, only elevated thyroid hormones turned out to be a predictor for response to sleep deprivation. PET and SPECT studies have convergently demonstrated an elevated metabolism in parts of the limbic system (e.g., the anterior cingulum) at baseline in responders. These findings do not yet allow conclusions with respect to the neurotransmitter systems involved.

Wiegand et al. (1993) investigated whether scheduled daytime naps can induce relapses after successful sleep deprivation therapy. The timing of the nap turned out to be a crucial factor; nap sleep duration and sleep structure during naps were less important.

The majority of studies in this field suffers from a methodological problem: there is no objective continuous polysomnographic measurement of sleep. The continuous absence of sleep during the sleep deprivation period is thus not documented. It is known from sleep deprivation studies in healthy probands that during prolonged sleep deprivation, short sleep episodes ("microsleep") occur frequently. Hemmeter et al. (1998) were the first to demonstrate that also in depressed patients undergoing sleep deprivation, microsleep occurs and tends to prevent the antidepressant effect. Data from a recently finished study of our group point into the same direction (partly published in Wiegand et al. 2002).

To further elucidate this question, an experimental procedure appears useful where the occurrence of sleep episodes during the sleep deprivation period is suppressed as far as possible by the vigilance enhancing drug modafinil.

The study aims to investigate whether the administration of modafinil or placebo during a 40 hour sleep deprivation period in depressed patients can intensify the antidepressant effect of the sleep deprivation.

This study is a basic science study that aims to provide information on the therapeutic mechanism of sleep deprivation in depression and on the reoccurence of depressive symptoms in case of intermittent short sleep episodes.

Primary Hypothesis:

There is a significant reduction on the HAMD-6 scale between baseline and 24 h later (at the mornings before and after one night of sleep deprivation)

Secondary Hypotheses:

1. The amount of "responders" (50% of reduction on the HAMD-6 scale) is significantly greater in the modafinil than in the placebo group.
2. The primary hypothesis and the first secondary hypothesis are also assessed by a self-rating scale of global mental state (Befindlichkeitsskala (Bf-s)) and by the Stanford Sleepiness Scale.
3. The overall amount of sleep assessed by polysomnography is smaller in the modafinil group as compared to the placebo group during the 40 h sleep deprivation period.
4. The group differences in HAMD-6 ratings are parralleled by differences in the overall amount of sleep during the 40 h sleep deprivation period.
5. There are group differences (Modafinil versus Placebo) on a comprehensive neuropsychological battery taken at baseline and 24 h later (at the mornings before and after one night of sleep deprivation)

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of the Psychiatric Hospital of the Technical University of Munich
* Diagnoses: Depressive episode with somatic symptoms (ICD-10: F32.01, F32.11, F32.21) or Recurrent depressive disorder with somatic symptoms (F33.01, F33.11, F33.21) or Bipolar affective disorder, presently depressive episode with somatic syndrome (F31.31, F31.41)
* Age 18 - 70 years
* Hamilton Depression Score (HAMD-21) at baseline > 18
* Women at child-bearing age have to provide a negative pregnancy test before study inclusion and have to use an effective, reliable and safe method of contraception throughout the study
* The patient must be able to understand the explanations about the study and to understand and follow the instructions of the investigator
* The patient is not involuntarily hospitalized under German law (§ 63 Strafgesetzbuch)

Exclusion Criteria:

* Presence of psychotic symptoms ICD-10: F32.3, F33.3, F31.5)
* Present psychiatric comorbidity (e.g. substance dependence)
* Relevant medical conditions
* Acute suicidality
* History of seizures
* Paroxysmal EEG activity
* Contraindications against treatment with modafinil (please see the most recent product information from August 2006:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Improvement on the Hamilton Depression Scale (6-Item Version) from Baseline to Follow-up | Baseline, 24 h (after sleep deprivation night), 48 h (after the first recovery night)

SECONDARY OUTCOMES:
Number of responders (50% reduction on the HAMD-6) in the modafinil group versus the placebo group | Baseline, 24 h (after sleep deprivation night), 48 h (after the first recovery night)
self-rating scale of global mental state (Befindlichkeitsskala (Bf-s)) and the Stanford Sleepiness Scale. | Baseline 24 h (after sleep deprivation night), 48 h (after the first recovery night)
Polysomnography (among others assessing sleep onset latency, sleep efficiency, sleep states, wakefulness after sleep onset) | Baseline 24 h (after sleep deprivation night), 48 h (after the first recovery night)
Neuropsychological battery (including Zahlenverbindungstest, California Verbal Learning Test, d2 Attention Stress Test, Farb-Wort-Interferenztest, CS fine motor task | Baseline 24 h (after sleep deprivation night), 48 h (after the first recovery night)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Wiegand, Prof. Dr.med. Dipl. Psych., Principal Investigator — Head of the Centre for Sleep Disorders
Locations (1):
- Centre for Sleep Disorders of the Department of Psychiatry and Psychotherapy, Munich, Germany

REFERENCES:
- [Background] Giedke H, Schwarzler F. Therapeutic use of sleep deprivation in depression. Sleep Med Rev. 2002 Oct;6(5):361-77. PMID 12531127
- [Background] Gillin JC, Buchsbaum M, Wu J, Clark C, Bunney W Jr. Sleep deprivation as a model experimental antidepressant treatment: findings from functional brain imaging. Depress Anxiety. 2001;14(1):37-49. doi: 10.1002/da.1045. PMID 11568981
- [Background] Hemmeter U, Bischof R, Hatzinger M, Seifritz E, Holsboer-Trachsler E. Microsleep during partial sleep deprivation in depression. Biol Psychiatry. 1998 Jun 1;43(11):829-39. doi: 10.1016/s0006-3223(97)00297-7. PMID 9611673
- [Background] Ringel BL, Szuba MP. Potential mechanisms of the sleep therapies for depression. Depress Anxiety. 2001;14(1):29-36. doi: 10.1002/da.1044. PMID 11568980
- [Background] Wirz-Justice A, Van den Hoofdakker RH. Sleep deprivation in depression: what do we know, where do we go? Biol Psychiatry. 1999 Aug 15;46(4):445-53. doi: 10.1016/s0006-3223(99)00125-0. PMID 10459393
- [Background] Wiegand M, Riemann D, Schreiber W, Lauer CJ, Berger M. Effect of morning and afternoon naps on mood after total sleep deprivation in patients with major depression. Biol Psychiatry. 1993 Mar 15;33(6):467-76. doi: 10.1016/0006-3223(93)90175-d. PMID 8490073
- [Background] Wu JC, Bunney WE. The biological basis of an antidepressant response to sleep deprivation and relapse: review and hypothesis. Am J Psychiatry. 1990 Jan;147(1):14-21. doi: 10.1176/ajp.147.1.14. PMID 2403471
- [Background] Kasper S, Möller HJ (eds). Therapeutischer Schlafentzug. Klinik und Wirkmechanismen. Wien New York: Springer, 1996
- [Background] Wiegand MH. Schlaf, Schlafentzug und Depression. Experimentelle Studien zum therapeutischen Schlafentzug. Berlin Heidelberg New York: Springer, 1995
- [Background] Wiegand MH, Jahn T, Schröder MM, Pohl C, Veselý B, Veselý Z, Brückner T, Bäuml J. Spontaneous sleep and microsleep episodes and mood in depressed patients during 40 hours of sleep deprivation therapy. Eur Arch Psychiat Clin Neurosci 256 Suppl. 2, II751, 2006